CLINICAL TRIAL: NCT02551835
Title: The Effect of Vitamin D Supplementation on Markers for Cardiovascular Disease and Diabetes: an Individual Participant Data Meta-analysis of Randomized Controlled Trials
Brief Title: Vitamin D Supplements on Markers for Cardiovascular Disease and Diabetes: an Individual Participant Data Meta-analysis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: European Union (Other)
Responsible Party: Principal Investigator, Karin Swart, PhD, Amsterdam UMC, location VUmc
Other Study IDs: ODIN 8.3
Record Dates: First submitted 2015-09-10; First posted 2015-09-16 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-03

CONDITIONS: Vitamin D Deficiency; Vitamin; Excess Vitamin D (Nutritional)
Keywords: ODIN; Meta-analysis; Cholecalciferol; 25(OH)D; Subgroup effects
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (12):
- Tromso Impaired Glucose Tolerance (IGT) study: RCT on 20000 IU vitamin D3/week versus placebo for 1 year among persons with impaired glucose tolerance and/or impaired fasting glucose.
- Tromso OBESITY study: RCT on 20000 or 40000 IU vitamin D3/week plus 500 mg calcium/day versus placebo plus 500 mg calcium/day for 1 year among persons with a high body mass index.
- Tromso Bone Mineral Density (BMD) study: RCT on 40000 IU vitamin D3/week plus 800 IU/day and 1000 mg calcium/day versus placebo plus 800 IU/day and 1000 mg calcium/day for 1 year among women with a low bone mineral density.
- Tromso CLAMP study: RCT on 40000 IU vitamin D3/week versus placebo for 6 months among persons with 25(OH)D values <42 nmol/L.
- Tromso DEPRESSION study: RCT on 40000 IU vitamin D3/week versus placebo for 6 months among persons with 25(OH)D values <55 nmol/L.
- Styrian Vitamin D Hypertension Trial: RCT on 2800 IU vitamin D3/day versus placebo for 8 weeks among persons a history of arterial hypertension and 25(OH)D values <75 nmol/L.
- Paravit study: RCT on 7000 IU vitamin D3/day versus placebo for 6 months among persons with a high body mass index and 25(OH)D values <50 nmol/L.
- Oosterwerff study: RCT on 1200 IU vitamin D3/day plus 500 mg calcium/day versus placebo plus 500 mg calcium/day for 16 weeks among non-western immigrants with pre-diabetes and 25(OH)D values <50 nmol/L.
- Chel study: RCT on 600 IU vitamin D3/day (or daily equivalent) versus placebo for 4 months among nursing home residents >70 years of age.
- Wicherts study: RCT on 800 IU vitamin D3/day versus 100,000 IU/3 months versus sunlight advice for 6 months among non-western immigrants with 25(OH)D values <25 nmol/L.
- University College Cork (UCC) 1 study: RCT on 200, 400, or 600 IU vitamin D3/day versus placebo for 22 weeks among persons > 63 years of age.
- UCC 2 study: RCT on 200, 400, or 600 IU vitamin D3/day versus placebo for 22 weeks among persons 20-40 years of age.

SUMMARY:
This meta-analysis will be conducted to study the effect on vitamin D supplements on markers for cardiovascular disease and diabetes using individual participant data from 12 RCTs. Given that previous data suggest that vitamin D supplementation might be most effective in those individuals with very low 25-hydroxyvitamin D (25(OH)D) and potentially harmful in those achieving very high levels after vitamin D supplementation, this meta-analyses will be performed in subgroups according 25(OH)D levels.

DETAILED DESCRIPTION:
Large randomized controlled trials (RCTs) are currently on-going to evaluate non-skeletal effects of vitamin D supplementation in the general older population. The results of these studies can be expected in 2017 to 2020 and while they will report important data, they may still leave knowledge gaps on the effects of vitamin D on clinically relevant surrogate parameters in specific groups. Recent data indicate that the association of vitamin D status and outcome is U- or reverse J-shaped and may be modified by the presence of certain risk factors or genetic variations of the vitamin D receptor.

This work is part of the European Union-project 'Food-based solutions for eradication of vitamin D deficiency and health promotion throughout the life cycle' (ODIN). This individual patient meta-analysis of existing high quality vitamin D RCTs aims to evaluate whether there are beneficial or harmful vitamin D effects on surrogate parameters for clinical outcomes (i.e. blood pressure, lipids, parathyroid hormone (PTH), fasting blood glucose and glycated haemoglobin (HbA1c)). With data from almost 3000 randomized subjects from 12 RCTs that are available within this consortium, the investigators will have sufficient power to detect clinically relevant effects of vitamin D supplementation on risk factors for cardiovascular disease.

Subgroup analyses will investigate effect modifiers to evaluate whether certain groups of individuals experience pronounced or attenuated effects from vitamin D supplementation. Given that previous data suggest that vitamin D supplementation might be most effective in those individuals with very low 25(OH)D and potentially harmful in those achieving very high levels after vitamin D supplementation, this individual patient data meta-analyses will be performed in subgroups with serum 25(OH)D levels <30, 40, and 50 nmol/L and >100, 125 and 150 nmol/L. 25(OH)D levels will be re-measured to ensure comparability.

ELIGIBILITY:
Inclusion Criteria:

* Availability of quality bio-banked samples for uniform 25(OH)D re-measurement
* Prospective data on one or more of the outcomes
* Willingness to collaborate

Exclusion Criteria:

* Trials among pregnant women, children, or performed in patient populations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participating RCTs are the Tromso IGT, Tromso OBESITY, Tromso BMD, Tromso CLAMP, Tromso DEPRESSION, Styrian Vitamin D Hypertension Trial, Paravit, Oosterwerff, Chel, Wicherts, UCC1, and UCC2 trials.
Sampling Method: Probability Sample
Enrollment: 2945 (Actual)
Dates: Start 2015-04; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | Participants were followed for the duration of the intervention period (range 8 weeks - 1 year, depending on the RCT in which they are participating)
  Systolic and diastolic (Main outcome of cardiovascular markers)
HbA1c | Participants were followed for the duration of the intervention period (range 8 weeks - 1 year, depending on the RCT in which they are participating)
  (Main outcome of diabetic markers)

SECONDARY OUTCOMES:
High-density lipoproteins (HDL) cholesterol | Participants were followed for the duration of the intervention period (range 8 weeks - 1 year, depending on the RCT in which they are participating)
Low-density lipoproteins (LDL) cholesterol | Participants were followed for the duration of the intervention period (range 8 weeks - 1 year, depending on the RCT in which they are participating)
Total cholesterol | Participants were followed for the duration of the intervention period (range 8 weeks - 1 year, depending on the RCT in which they are participating)
Triglycerides | Participants were followed for the duration of the intervention period (range 8 weeks - 1 year, depending on the RCT in which they are participating)
Parathyroid hormone (PTH) | Participants were followed for the duration of the intervention period (range 8 weeks - 1 year, depending on the RCT in which they are participating)
  Parathyroid hormone
Fasting glucose | Participants were followed for the duration of the intervention period (range 8 weeks - 1 year, depending on the RCT in which they are participating)
Fasting insulin | Participants were followed for the duration of the intervention period (range 8 weeks - 1 year, depending on the RCT in which they are participating)
C-peptide | Participants were followed for the duration of the intervention period (range 8 weeks - 1 year, depending on the RCT in which they are participating)
Two-hour glucose | Participants were followed for the duration of the intervention period (range 8 weeks - 1 year, depending on the RCT in which they are participating)
  After oral glucose tolerance test

REFERENCES:
- [Derived] Swart KM, Lips P, Brouwer IA, Jorde R, Heymans MW, Grimnes G, Grubler MR, Gaksch M, Tomaschitz A, Pilz S, Eiriksdottir G, Gudnason V, Wamberg L, Rejnmark L, Sempos CT, Durazo-Arvizu RA, Dowling KG, Hull G, Skrabakova Z, Kiely M, Cashman KD, van Schoor NM. Effects of vitamin D supplementation on markers for cardiovascular disease and type 2 diabetes: an individual participant data meta-analysis of randomized controlled trials. Am J Clin Nutr. 2018 Jun 1;107(6):1043-1053. doi: 10.1093/ajcn/nqy078. PMID 29868916